CLINICAL TRIAL: NCT05617066
Title: Psychological Stress and Systemic Sclerosis
Brief Title: Stress, Scleroderma and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asociación Española de Esclerodermia (Other)
Responsible Party: Principal Investigator, Eva Montero Lopez, Principal investigator. PhD in Psychology. Clinic Psychologist, Asociación Española de Esclerodermia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: AEE
Record Dates: First submitted 2022-11-09; First posted 2022-11-15 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Scleroderma
Keywords: scleroderma, stress, cognitive behavioral therapy
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- therapy vs psychological support and usual care (Active Comparator): Comparison between therapy groups vs psychological support and usual care. Only one group receive therapy.
  Interventions: Behavioral: Cognitive behavioral therapy
- therapy and psychological support versus control group (No Intervention): Comparison between therapy groups vs psychological support and usual care. Only one group receive therapy.

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — With the cognitive behavioral therapy will work on different aspects for coping and tools psychological stress.
  Arms: therapy vs psychological support and usual care

SUMMARY:
150 patients of legal age will participate in this project, diagnosed with systemic sclerosis.

Patients will be randomly assigned, as will be detailed later, to one of the following three groups:

Therapy Group (GT): This group will be made up of 50 patients who will receive cognitive behavioral therapy of coping with stress (online modality) in groups of 10-12 people during twelve sessions Consecutive weekly courses of 1.5 to 2 hours duration taught by psychology professionals. of this mode 4 subgroups will be made. Psychological Support Group (AP): This group will be made up of 50 patients who will receive psychoeducation about stress and its consequences and the specific stress suffered by people with a autoimmune disease such as scleroderma. It will have a duration of twelve weekly sessions.

Consecutive sessions of 1.5 to 2 hours in length taught by professional psychologists. In this way they will 4 subgroups. Usual Care Group (CG): This group will be made up of 50 patients who will follow their usual care. Later, once the study is over, they will be offered to participate in coping with stress to the person who is interested.

DETAILED DESCRIPTION:
150 elderly patients diagnosed with systemic sclerosis in any of its variants, both diffuse, limited or sine scleroderma.

The inclusion criteria are: diagnosis made by a medical specialist, good command of the Spanish language (oral and written comprehension) and have an internet connection. As exclusion criteria they must not suffer no psychiatric illness. Patients will be randomly assigned into each of the three groups.

Informed consent. Patients must be informed in writing of the objectives of the project and of the work protocol in which they are going to be included. Once read and understood, They will sign the consent. The research staff is obliged to save said consents.

Confidentiality and data protection commitment. Ethical principles will be followed and deontological related to psychological research collected in the main codes currently nationally or internationally: The Code of the Official College of Psychologists (1987), the Meta- Code of the European Federation of Psychological Associations (1995), and The Ethical Principles and Code of Conduct of Psychologists of the American Psychological Association (2002).

Instruments:

All the evaluation as well as the therapies will be carried out online through Google Form and GoogleMeet, where questions regarding sociodemographic variables and information will be asked related to variables about your disease: disease variant (ESd, ESl or ESss), profile of autoantibodies, age at diagnosis, evolution time, presence of Raynaud's, current digital ulcers, pulmonary hypertension, interstitial lung disease, esophageal involvement, intestinal involvement, renal or cardiac involvement; as well as current treatment. Information will also be collected on possible comorbidities: high blood pressure, diabetes, hypercholesterolemia or hypertriglyceridemia, and toxic habits such as tobacco and/or alcohol use.

For the psychological evaluation, the following instruments will be completed:Perceived Stress Scale (EEP-14). It's about a instrument that evaluates the perception of stress in different life situations. It is composed of fourteen items on a five-point Likert-type scale. It has adequate reliability (consistency internal=.81 and test-retest= 0.73). Stress Vulnerability Inventory (IVE). This questionnaire assesses the individual's predisposition to be influenced by perceived stress. This composed of twenty-two dichotomous items and the maximum value that can be obtained is twenty-two points. The Cronbach's alpha reliability coefficient is 0.87.

Connor and Davidson Resilience. Assesses resilience being understood as the individual's ability to coping and adapting to circumstances, is made up of twenty-five Likert-type scale items of five points; higher scores reflect greater resilience. It has good reliability with an alpha of Cronbach of 0.89. Revised Symptom Inventory (SCL-90-R). It is an instrument with ninety items on a five-point Likert-type scale, zero being nothing and four much, which evaluates nine dimensions: somatization, obsession-compulsion, depression, anxiety, hostility, phobic anxiety, paranoid ideation and psychoticism. The scale also consists of seven extra items distributed into three global distress indices: the GSI, which measures global psychological distress, the PSDI, which is used to measure the intensity of symptoms and the Total Symptom Index which is used to measure the number of symptoms that the person reports. The scores are transformed into percentiles (0-100), in this line the percentiles ≥75 represent clinical symptoms in any of the subscales of this instrument. The nine dimensions show acceptable reliability, with Cronbach's alpha for internal consistency of 0.81.

EUROQOL-5Q health questionnaire. Measure quality of life related to health (HRQoL) both in the general population and in groups of patients with different pathologies. The individual himself assesses his state of health, first in levels of severity by dimensions and then on a more general assessment visual analog scale. A third element is the index of values that is obtained for each state of health generated by the instrument. The descriptive system contains five dimensions of health (mobility, self-care, activities of daily living, pain/discomfort, and anxiety/depression) and each of them has three levels of severity (no problems, some problems or moderate problems and serious problems). In this part of the questionnaire the individual must mark the level gravity corresponding to his state of health in each of the dimensions, referring to the same day to complete the questionnaire. In each dimension, severity levels are coded 1 if the response option is "no (I have) problems"; with a 2 if the answer option is "some or moderate problems"; and with a 3 if the answer option is "many problems".

DIENER life satisfaction scale.It consists of five items that assess satisfaction with life through the global judgment that people make about this from the degree of agreement (from 1: STRONGLY DISAGREE to 5: STRONGLY AGREE) on five aspects: if the type of life is similar to what has always been dreamed of having, if the conditions of life are excellent, if I am satisfied with my life, if important things have been obtained and finally if I could live again I would like everything to be the same.

Short Survey on Health SF-36.Short survey on health of 36 items (SF-36) of. The 36 items measure eight dimensions: Physical function (limitations in physical activities due to health problems), Social function (limitations in social activities due to physical or emotional problems), Physical role (limitations in activities of roles due to physical health problems), Body pain, General mental health (discomfort and well-being), Social Role (limitations in usual role activities due to problems emotional), Vitality (energy and fatigue), Perception of general health.

Evaluation of cortisol concentrations in hair: Strands of hair with a diameter of Approximately 3 mm, near the scalp, in the middle posterior region of the head, where the has indicated less variability in cortisol levels. They will be cut with scissors clean as close to the scalp as possible, not including the hair follicle itself, not recommended for analysis. Each hair sample will be kept in aluminum foil and inside an airtight bag, so that neither light nor moisture penetrates the sample. For this, each participant will be sent both a tutorial as an envelope with the entire kit for collecting and storing the sample (except the scissors), for once collected, they are sent to the laboratory of the Faculty of Pharmacy of the University of Granada, where the levels of cortisol in hair will be analyzed and obtained. This whole process will be totally free for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis made by a specialist doctor, good command of the Spanish language (oral and written comprehension) and have an internet connection.

Exclusion Criteria:

* No psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-11-26 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Cortisol y psychological stress levels | 3 months
  Decreased cortisol and psychological stress after therapy

SECONDARY OUTCOMES:
Quality of life and psychological status | 3 months
  Improvement of quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No